CLINICAL TRIAL: NCT00315913
Title: Placebo-Controlled Randomized Trial of Oxytocin Alone Versus Oxytocin and Propranolol for the Treatment of Dysfunctional Labor
Brief Title: Trial of Oxytocin Alone Versus Oxytocin and Propranolol for the Treatment of Abnormal Labor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Deborah A. Wing, Professor and MFM Division Director, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS #2004-3997
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Dysfunctional Labor
Keywords: Labor; Dysfunctional Labor; Labor Arrest; Primary Cesarean Section Prevention
MeSH Terms: conditions — Dystocia | interventions — Propranolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Propranolol (Experimental): IV dose propranolol
  Interventions: Drug: Propranolol
- IV Placebo (Placebo Comparator): IV Placebo of saline solution equal to propranolol in volume
  Interventions: Other: IV Placebo

INTERVENTIONS:
Drug: Propranolol — IV Propranolol 1mg/min for a total of 2 minutes. Total dose 2mg
  Other Names: Inderal
  Arms: IV Propranolol
Other: IV Placebo — IV Saline Solution
  Other Names: Normal Saline
  Arms: IV Placebo

SUMMARY:
The purpose of this study is to determine whether propranolol is better than oxytocin for the treatment of labor abnormalities. The endpoint is the rate of vaginal delivery experienced by women receiving prolonged oxytocin versus propranolol.

DETAILED DESCRIPTION:
This trial was designed to test if propranolo can reduce the c section rate for dysfuctional labor. Due to stringent inclution and exclusion criteria and low enrollment the study was closed.

ELIGIBILITY:
Inclusion Criteria:

* Must be term pregnancy (> 37 weeks)
* Vertex presentation
* Active labor (4-5 centimeters dilated)

Exclusion Criteria:

* Heart disease
* Diabetes
* Currently taking propranolol
* Contraindications to labor or vaginal delivery
* Multiple gestations
* Preterm
* Chorioamnionitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Battista, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States